CLINICAL TRIAL: NCT00904930
Title: Evaluation of the Periotest Method as a Tool for Tooth Mobility Monitoring and Splint Rigidity Assessment in Dental Traumatology
Brief Title: Evaluation of the Periotest Method in Dental Traumatology
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Other Study IDs: PT-WCS1-WCS2-Hu
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Dental Trauma
Keywords: Tooth mobility assessment; Splinting; Splint Rigidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no periodontal disease: 33 dental students (13 male, 20 female) with a mean age of 24.7 years (min. 19.8; max. 36.5) with no periodontal disease or dental trauma
  Interventions: Device: Wire Composite Splint (Dentaflex 0.45 mm); Device: Wire Composite Splint (Denture Strengtheners)

INTERVENTIONS:
Device: Wire Composite Splint (Dentaflex 0.45 mm) — Wire-Composite-Splint: Dentaflex 0.45 mm (Dentaurum, Pforzheim, Germany) attached with Tetric flow (IvoclarVivadent, Schaadn, Liechtenstein) to the teeth
Device: Wire Composite Splint (Denture Strengtheners) — Wire-Composite-Splint: Denture Strengtheners 0.8x1.8 mm (Dentaurum, Pforzheim, Germany) attached with Tetric flow to the teeth

SUMMARY:
Background/Aims: The Periotest® method represents a technique for objective tooth mobility assessment. The aims of this study were: 1. receiving information about normal Periotest® values in vertical and horizontal dimension on periodontally healthy teeth for individuals aged 20-35, 2. investigating the reliability of the Periotest® method in terms of intra-serial and inter-serial reproducibility before splinting and with an applied dental trauma splint, 3. evaluating the splint effect of two different wire-composite splints in vivo.

Materials and Methods: On periodontally healthy dental students (n=33; mean age 24.7 years) Periotest® values were measured on reproducible measuring points, in vertical and horizontal dimension and before splinting and after splint insertion. Three readings were taken per serial to observe the intra-serial reproducibility, and for testing inter-serial reproducibility three serials were measured (Friedman-test; P ≤ 0.001). Two different wire-composite-splints (1 = Dentaflex 0.45 mm, 2 = Strengtheners 0.8x1.8) were inserted, the Periotest® values were measured and the splint effects were calculated and compared (Whitney-Mann-U-test; P ≤ 0.001).

ELIGIBILITY:
Inclusion Criteria:

* age 19-36
* healthy upper front teeth

Exclusion Criteria:

* periodontal disease
* orthodontic treatment during the investigation period
* history of dental trauma
* fillings or restorations on upper front teeth
* endodontically treated teeth

Ages: 19 Years to 36 Years | Sex: All
Age Groups: Adult
Study Population: Dental students Dental Clinic 1 and 2
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Bavaria, Germany